CLINICAL TRIAL: NCT01161186
Title: A Phase I Study of Nab-paclitaxel (Abraxane), Gemcitabine, and Capecitabine (Xeloda) (AGX) in Patients With Previously Untreated, Metastatic Pancreatic Adenocarcinoma
Brief Title: Nab-paclitaxel (Abraxane), Gemcitabine, and Capecitabine (Xeloda) for Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC#10451
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Pancreatic Neoplasms; Pancreatic Cancer; Adenocarcinoma
Keywords: pancreas; cancer; abraxane; metastatic; gemcitabine; capecitabine; adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Neoplasms; Neoplasm Metastasis | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Capecitabine; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nab-paclitaxel,Gemcitabine, and Capecitabine (Experimental)
  Interventions: Drug: nab-paclitaxel, gemcitabine, capecitabine

INTERVENTIONS:
Drug: nab-paclitaxel, gemcitabine, capecitabine — {nab-paclitaxel: Intravenous, 100 to 150 mg/m2 over 30 minutes once per cycle.} {gemcitabine: Intravenous, 750 to 1000 mg/m2 at 10mg/m2/minute once per cycle.} {capecitabine: oral, 500 to 1000 mg/m2 b.i.d. 7 days per cycle}
  Other Names: Abraxane; nanoparticle albumin bound paclitaxel; Xeloda; Gemzar

SUMMARY:
The purpose of this study is to evaluate optimal dose and safety of the combination of Abraxane, gemcitabine, and Xeloda (capecitabine) (AGX) as first-line therapy in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma (PDAC) represents the fourth leading cause of cancer-related mortality in the United States, with an estimated 35,240 deaths attributable to PDAC in 2009 (1). Over 90% of patients have inoperable disease at presentation, at which point systemic therapy becomes the primary form of treatment. Single agent gemcitabine became the standard of care for advanced pancreatic cancer a decade ago since demonstrating improved survival when compared with fluorouracil. Since then, a number of phase III trials have evaluated the benefit of adding additional cytotoxic or targeted agents to gemcitabine (2-17).

The PA.3 trial (15), which led to the approval of erlotinib in advanced pancreatic cancer, was a landmark study in that it represented the first positive phase III study of a combination regimen for this disease indication; however, while erlotinib represents both an important proof of principle and a welcome addition to our therapeutic armamentarium, it has failed to gain significant traction in this disease, as many in the oncology community consider the marginal absolute improvement in median overall survival to be of questionable clinical significance.

While these studies individually have failed to consistently demonstrate a survival advantage for gemcitabine-based combination therapy, a recent meta-analysis did show that the addition of either a platinum analog or a fluoropyrimidine to gemcitabine does result in a significant improvement in overall survival compared to gemcitabine alone, particularly in patients with a preserved performance status (18). As described in the following section, the combination of gemcitabine and capecitabine may be a particularly attractive cytotoxic doublet to build upon.

Gemcitabine/capecitabine for pancreatic cancer

Gemcitabine and capecitabine have demonstrated synergy in pre-clinical studies, thought to be due to several mechanisms. Capecitabine is converted to fluorouracil in tissues by pyrimidine nucleoside phosphorylase (PyNPase), which is over-expressed in many tumors (19). In breast cancer xenograft models, gemcitabine has been shown to cause increased expression of PyNPase, which may in turn enhance the conversion of capecitabine to 5-FU (20). An intermediate of gemcitabine also leads to enhanced binding of the active metabolite of 5-FU to thymidylate synthase, further augmenting the action of capecitabine (21).

Preliminary analysis of one of these studies did show a significant survival benefit with the combination arm (overall survival 7.4 months versus 6 months; 1 year survival 26% versus 19%); however, final data from this trial have not yet been published (3). A subsequent phase III Swiss trial did not demonstrate a significant improvement in overall survival with the combination of gemcitabine/capecitabine as compared to gemcitabine alone; however, a subset analysis in patients with good performance status (KPS 90-100) did show a significant survival improvement from 7.4 months to 10.1 months in those who received the combination regimen (4).

Several strategies may further optimize the dose, schedule, and administration of both gemcitabine and capecitabine. First, delivery of gemcitabine at a fixed-dose rate infusion (FDR) (10 mg/m2/min) maximizes the intracellular accumulation of the triphosphate form of this drug. This approach has been evaluated in both a randomized phase II and a phase III cooperative group trial (ECOG 6201), with some suggestion of benefit compared to standard-infusion gemcitabine given over 30 minutes (9, 22). Second, administering capecitabine in a biweekly fashion (7 days on followed by 7 days off) rather than in the standard 2-week on, 1-week off fashion may allow for dose intensification without increasing toxicity (23, 24) (see also Part E. below).

The GTX Regimen

The addition of a taxane to gemcitabine/capecitabine has previously been evaluated in the so-called GTX regimen (fixed-dose rate gemcitabine, docetaxel, capecitabine) (26). Studies of GTX in advanced pancreatic cancer patients (26, 27) and locally advanced unresectable disease (28) have revealed encouraging efficacy data.

Abraxane (nab-paclitaxel)

Abraxane (nab-paclitaxel, nanoparticle albumin-bound paclitaxel; formerly ABI-007) is a Cremophor® EL-free, albumin-bound form of paclitaxel with a mean particle size of approximately 130 nanometers. This composition provides a novel approach of increasing intra-tumoral concentrations of the drug by a receptor-mediated transport process allowing transcytosis across the endothelial cell.

Preclinical studies comparing Abraxane to Taxol (paclitaxel Cremophor EL solvent-based, BMS) demonstrated lower toxicities, with an MTD approximately 50% higher for Abraxane compared to Taxol. At equal doses there was less myelosuppression and improved efficacy in a xenograft tumor model of human mammary adenocarcinoma. At equitoxic doses of paclitaxel, Abraxane was found to be markedly more efficacious than Taxol (29).

The current FDA-approved indication of Abraxane is for the treatment of breast cancer after failure of combination chemotherapy for metastatic disease or relapse within 6 months of adjuvant chemotherapy (prior therapy should have included an anthracycline unless clinically contraindicated).

Our choice of nab-paclitaxel for this proposal is based on provocative preclinical and clinical data suggesting efficacy of the agent in pancreatic cancer. Specifically, binding of nab-paclitaxel by an albumin specific receptor (gp60) leads to subsequent activation of a protein caveolin-1, which mediates internalization of the compound into the endothelial cell and transport through the bloodstream to the tumor interstitium. SPARC (Secreted Protein And Rich in Cysteine), a tumor-secreted protein, binds albumin, releasing the active drug at the tumor cell membrane, thereby increasing its concentration at the target site of action. SPARC is known to be over-expressed in pancreatic cancers, leading to an interest in studying nab-paclitaxel in this disease.

The combination of nab-paclitaxel and gemcitabine in advanced pancreatic cancer demonstrated very promising results in a phase I/II study (31). In that study, the maximum tolerated dose of nab-paclitaxel when given concurrently with gemcitabine was 125 mg/m2, both agents administered weekly x 3 of 4. This same combination of nab-paclitaxel (125 mg/m2) and gemcitabine (1000 mg/m2) was also shown to be well tolerated in a phase II trial in metastatic breast cancer (32), with both agents administered on a 2-week-on, 1-week-off schedule. Of note, the pivotal study upon which nab-paclitaxel was approved for use in breast cancer used a dose of 260 mg/m2, as a single agent, on an every 3 week schedule.

The doses of nab-paclitaxel to be tested in our proposed dose-escalation trial, when combined with gemcitabine and capecitabine using an alternating-week dose schedule, will range between 75 and 150 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed pancreatic adenocarcinoma
2. Stage IV disease (metastatic only)
3. No prior systemic therapy for their diagnosis (except in adjuvant setting > six months previously)
4. ECOG performance score of 0-1
5. At least 18 years of age
6. Evidence of either or both of the following:

   * RECIST-defined measurable disease (lesions that can be accurately measured in at least one dimension with the longest diameter ≥ 20mm using conventional techniques or ≥10 mm with spiral CT scan)
   * An elevated serum CA19-9 at baseline ( ≥ 2X ULN)
7. Female patients must be either surgically sterile or postmenopausal, or if of childbearing potential must have a negative pregnancy test (serum or urine) prior to enrollment and agree to use effective barrier contraception during the period of therapy. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the investigator.
8. Adequate bone marrow function:

   * ANC ≥ 1500/uL
   * platelet count ≥ 100,000/uL
   * hemoglobin ≥ 9.0 g/dL
   * Total bilirubin ≤ 1.5 X ULN
   * AST (SGOT) ≤ 2.5 X ULN
   * ALT (SGPT) ≤ 2.5 X ULN

10. Adequate renal function as determined by either:

* Calculated or measured creatinine clearance ≥ 40 mL/min (for calculated creatinine clearance, Cockroft-Gault equation will be used). The Modified Cockcroft-Gault formula is as follows:

((140 - age(yrs)) x (actual weight(kg))) / (72 x serum creatinine(mg/dl))

* Multiply by another factor of 0.85 if female
* Serum creatinine ≤ 1.5 X ULN 11. Ability to swallow oral medications 12. Ability to understand the nature of this study protocol and give written informed consent 13. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Any prior systemic or investigational therapy for metastatic pancreatic cancer. Systemic therapy administered alone or in combination with radiation in the adjuvant setting is permissible as long as it was completed > 6 months prior to the time of study enrollment.
2. Inability to comply with study and/or follow-up procedures.
3. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that, in the opinion of the investigator, renders the subject at high risk from treatment complications or might affect the interpretation of the results of the study.
4. Presence of central nervous system or brain metastases.
5. Life expectancy < 12 weeks
6. Pregnancy (positive pregnancy test) or lactation.
7. Prior malignancy except for adequately treated basal cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other form of cancer from which the patient has been disease-free for 5 years.
8. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
9. Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome.
10. Known, existing uncontrolled coagulopathy.
11. Pre-existing sensory neuropathy > grade 1.
12. Major surgery within 4 weeks of the start of study treatment, without complete recovery.
13. Concurrent/pre-existing use of coumadin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
to establish the maximal tolerated dose (MTD) of the AGX combination in patients with previously untreated, metastatic pancreatic adenocarcinoma. | Ongoing evaluation through sequential dose cohorts

SECONDARY OUTCOMES:
To assess the safety profile of this combination (AGX) using NCI-CTCAE v.4 criteria. | Ongoing evaluation for all patients throughout the course of treatment
To obtain a preliminary assessment of the clinical efficacy of AGX as measured by time to tumor progression, overall survival, objective radiographic response (ORR), and CA 19-9 biomarker response | Efficacy evaluations at 2-month intervals; patients followed for survival throughout lifetime.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ko, M.D., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Huntsman Cancer Institute, Salt Lake City, Utah